CLINICAL TRIAL: NCT03084965
Title: Retrospective Study of Patients With Type 2 Diabetes Mellitus on Dapagliflozin Therapy in Taiwan
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D1690R00022
Record Dates: First submitted 2017-03-15; First posted 2017-03-21 (Actual); Last update posted 2019-02-26 (Actual); Status verified 2019-02

CONDITIONS: Type II Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Retrospective Study of Patients With Type 2 Diabetes Mellitus on Dapagliflozin Therapy in Taiwan.

ELIGIBILITY:
Inclusion Criteria:

1. Outpatient equal to or more than 20 years of age.
2. T2DM patient initiated dapagliflozin after May 1st 2016 as a second line or third line oral anti-diabetic therapy, either as add-on or switching from one to another. Or initiating dapagliflozin as adjunctive therapy for T2DM subjects treated with insulin.
3. Completed follow-up of at least 6 months regardless of continuation on dapagliflozin therapy.
4. Will provide completed and signed written informed consents.

Exclusion Criteria:

1. Subjects with a history of SGLT2 inhibitor therapy other than dapagliflozin prior to Baseline.
2. Subjects with Type 1 diabetes.
3. Treatment with other investigational drugs concurrently during the retrospective data collection period.

Max Age: 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Type 2 Diabetes Mellitus patients on Dapagliflozin Therapy in Taiwan
Sampling Method: Non-Probability Sample
Enrollment: 1987 (Actual)
Dates: Start 2017-05-12 (Actual); Primary Completion 2018-03-02 (Actual); Study Completion 2018-03-02 (Actual)

PRIMARY OUTCOMES:
Change in HbA1c | 6 months
  To assess the change from baseline (time to initiate dapagliflozin*) in HbA1c at 6 months

CONTACTS AND LOCATIONS:
Locations (8):
- Taiwan (8):
  - Research Site, Changhua
  - Research Site, Chiayi City
  - Research Site, Kaohsiung City
  - Research Site, New Taipei City
  - Research Site, Taichung
  - Research Site, Tainan
  - Research Site, Taipei
  - Research Site, Taoyuan District

REFERENCES:
- See also: D1690R00022 Study Report Synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=14656&filename=D1690R00022_Study_Report_Synopsis.PDF